CLINICAL TRIAL: NCT01218360
Title: Observational Study on Disease Severity, Evaluation Tools and the Long Term Impact of Each Treatment Strategy in the Daily Clinical Practice in Patients With Moderate to Severe Active Crohn's Disease (Protocol P06484)
Brief Title: Observational Study of Disease Severity in Participants Diagnosed With Crohn's Disease and Long Term Impact of Treatment Strategies in Participants With Moderate to Severe Crohn's Disease (Protocol P06484)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P06484
Record Dates: First submitted 2010-10-07; First posted 2010-10-11 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Crohn Disease
Keywords: Crohn's disease; standard-of-care; Crohn Disease; Active Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants: All participants enrolled
  Interventions: Drug: Physician standard-of-care

INTERVENTIONS:
Drug: Physician standard-of-care — Participants will be treated according to their physician's routine practice and the respective Summary of Product Characteristics (SmPC).

SUMMARY:
This is an observational study to determine the prevalence of moderate to severe Crohn's disease (CD) among patients with active CD and to evaluate existing therapeutic trends in a standard clinical practice.

ELIGIBILITY:
Inclusion Criteria

1. Must have a diagnosis of active Crohn's Disease irrespective of severity,
2. Must be inadequately controlled with their current therapy and for whom physician

   decides to switch treatment.
3. Must be between 18 and 65 years of age, of either sex,
4. Must demonstrate willingness to participate in the study by signing the written informed consent.

Exclusion Criteria

* No specific exclusion criteria will be applied to a participant as long as the participant is eligible for the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with diagnosed active Crohn's Disease who are inadequately controlled with their current therapy
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2011-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Crohn's disease participants among the study population with a Crohn's Disease Activity Index (CDAI) score of 220-450 at the enrollment to the study. | Week 0
Record of treatment strategy followed | Week 0 to 2 years
Change in the CDAI score during the observational period | Week 0 to 2 years

SECONDARY OUTCOMES:
Number of surgeries and hospitalizations during the observational period | Week 0 to 2 years